CLINICAL TRIAL: NCT07405840
Title: Application of Autologous Stem Cells From Adipose Tissue in the Regeneration of Knee Joint Cartilage
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Clinical Center of Vojvodina (Other)
Responsible Party: Principal Investigator, Sasa Karan, Sasa Karan, MD, Orthopedic surgeon and Traumatologist, Clinical Center of Vojvodina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00-421/2024
Record Dates: First submitted 2026-01-22; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Osteearthritis
Keywords: osteoarthritis; stromal vascular fraction; chondroprotectors; regenerative orthopedic surgery
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SVF group (Experimental): In this arm, we included patients which will be treated with intraarticular injection of SVF from fat pad
  Interventions: Biological: stromal vascular fraction (SVF)
- CP group (Active Comparator): In this arm we will included patient swhich will be treated with Reviscon Re cross HA injection by MV Pharm
  Interventions: Drug: CP

INTERVENTIONS:
Biological: stromal vascular fraction (SVF) — Participants will undergo autologous adipose tissue harvesting under local anesthesia. The adipose tissue (1-5 mL) will be processed using the Lipocube® mechanical closed system to isolate stromal vascular fraction (SVF), containing adipose-derived stem cells (ADSCs), pericytes, and regenerative stromal cells. The prepared SVF will be injected intra-articularly into the affected knee under sterile conditions.
  Other Names: SVF
  Arms: SVF group
Drug: CP — Participants will receive a single intra-articular injection of high-molecular-weight hyaluronic acid (Reviscon Re-Cross, MV Pharm; 88 mg sodium hyaluronate [2.2%] in 4 mL solution) under sterile conditions.
  Arms: CP group

SUMMARY:
This randomized, controlled clinical trial will evaluate the safety and effectiveness of autologous adipose-derived stromal vascular fraction (SVF) therapy in patients with knee osteoarthritis (OA) grades II-IV, compared with standard chondroprotective (CP) treatment. The study will enroll male and female patients and follow them for 12 months, assessing pain (VAS), function (WOMAC, KOOS, SF-36), radiologic progression, and safety (adverse events). The trial aims to determine whether SVF therapy provides superior clinical outcomes and to inform evidence-based recommendations for OA management in the Serbian population.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a progressive degenerative joint disorder characterized by cartilage loss, subchondral bone remodeling, synovial inflammation, and joint pain. It is a leading cause of disability worldwide, particularly affecting weight-bearing joints such as the knee. The pathological process involves a combination of mechanical stress, inflammatory cytokine activity, and abnormal tissue remodeling, leading to progressive cartilage degradation and functional impairment. OA is increasingly recognized as a biologically active disease rather than a simple "wear-and-tear" condition, with complex interactions among chondrocytes, synoviocytes, immune cells, and extracellular matrix components.

Current non-surgical therapies, including analgesics, physiotherapy, and chondroprotective agents, primarily address symptom control and functional preservation, without altering the underlying degenerative process. Surgical interventions, such as osteotomy or total knee arthroplasty, are reserved for advanced disease but are associated with risks and limited applicability in younger or active patients. These limitations have prompted the exploration of regenerative medicine approaches that aim to restore joint homeostasis and promote cartilage repair.

Autologous adipose-derived stromal vascular fraction (SVF) has emerged as a promising regenerative therapy for knee OA. SVF is a heterogeneous cell population derived from adipose tissue, comprising mesenchymal stem cells (MSCs), pericytes, endothelial progenitors, and other stromal cells. These cells possess anti-inflammatory, immunomodulatory, and trophic properties that can support tissue repair both directly and indirectly. SVF may contribute to cartilage regeneration through differentiation of MSCs into chondrocytes, secretion of growth factors and cytokines that stimulate resident chondrocytes, modulation of synovial inflammation, and promotion of angiogenesis in the subchondral bone. Compared to bone marrow-derived MSCs, adipose tissue provides a more abundant and easily accessible source of regenerative cells with minimal donor site morbidity.

Preclinical studies and early clinical trials have demonstrated that intra-articular injection of adipose-derived SVF is feasible, safe, and associated with improvements in pain, function, and cartilage quality. However, there is a paucity of controlled clinical data directly comparing SVF therapy with standard chondroprotective interventions, particularly in the Serbian population. The present study is designed to address this gap by systematically evaluating the clinical efficacy, safety, and regenerative potential of SVF in patients with moderate to severe knee OA.

This trial will employ rigorous, standardized methodologies for SVF isolation and administration, using a closed mechanical system to obtain a highly viable and potent cell population. By combining clinical assessments with imaging-based evaluation of cartilage repair, this study aims to generate comprehensive data on both symptomatic and structural outcomes. The results are expected to provide critical evidence to support the integration of SVF therapy into standard orthopedic practice, potentially offering a regenerative alternative for patients with degenerative knee disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years).
* Radiologically confirmed knee OA (grades II-IV, Kellgren-Lawrence scale).
* KOOS pain score ≤ 60 points.
* Symptomatic degenerative knee disease with at least 6 months of persistent pain.
* No history of major knee trauma or prolonged immobilization (>10 days)

Exclusion Criteria:

* Minors (<18 years).
* Asymptomatic OA (KL grade 0-I).
* Severe axial deformity (varus >10°, valgus >10°).
* Current anticoagulant or antiplatelet therapy.
* Intra-articular corticosteroid injection within the past 6 months.
* History of major knee trauma or surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, 3 6 and 12 months post-treatment.
  Description: The WOMAC is a validated self-administered questionnaire measuring pain, stiffness, and physical function in patients with knee osteoarthritis. Each subscale is scored, with higher scores indicating greater disability.
  Purpose: To assess changes in pain, joint stiffness, and functional impairment over time.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline (pre-treatment) 3, 6 and 12 months post-intervention.
  Description: The KOOS is a patient-reported questionnaire assessing knee-related pain, symptoms, function in daily living, function in sports and recreation, and knee-related quality of life. Scores range from 0 (extreme problems) to 100 (no problems).Purpose: To evaluate overall knee function and symptom improvement following SVF or chondroprotective therapy.
Lysholm Knee Scoring Scale | Timepoints: Baseline, 3, 6 and 12 months post-treatment.
  Description: The Lysholm score evaluates knee function based on symptoms such as limp, support, locking, instability, pain, swelling, stair climbing, and squatting. Scores range from 0 (worst function) to 100 (normal function).
  Purpose: To quantify functional recovery and symptom improvement in daily activities.
Visual Analog Scale (VAS) for Pain | Baseline, 3,6 and 12 months post-treatment.
  Description: The VAS is a 100 mm scale where patients indicate their perceived pain intensity, from 0 (no pain) to 100 (worst possible pain).Purpose: To measure changes in subjective knee pain intensity over time.
MRI-based Cartilage Evaluation (MOCART Score) | Baseline and 12 months post-treatment.
  Description: The Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) score evaluates structural cartilage repair by assessing defect fill, integration to border zone, surface, structure, signal intensity, subchondral lamina, subchondral bone, adhesions, and synovitis. Scores range from 0 (worst repair) to 100 (optimal repair).
  Purpose: To assess morphological cartilage regeneration following intervention.
Short Form Health Survey (SF-36) | Baseline and 12 months post-treatment.
  Description: The SF-36 is a patient-reported survey evaluating health-related quality of life across eight domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional health, and mental health. Scores are transformed to a 0-100 scale, with higher scores indicating better health.
  Purpose: To assess changes in overall health-related quality of life after treatment.
Documentation of Adverse Events | Throughout the 12-month follow-up.
  Description: All local or systemic adverse events, including injection site reactions, swelling, pain exacerbation, infection, or other unexpected clinical events, will be recorded and categorized according to severity, duration, and relationship to the study intervention.
  Purpose: To evaluate the safety profile of SVF and standard chondroprotective therapies.

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Center of Vojvodina, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Garza JR, et al. Clinical efficacy of intra-articular mesenchymal stromal cells for the treatment of knee osteoarthritis: a double-blinded prospective randomized controlled clinical trial. Am J Sports Med. 2020;48(3):588-98.